CLINICAL TRIAL: NCT07110012
Title: The Role of Simulation-based Training in Resident Curriculum in Anaesthesia and Intensive Care
Acronym: STRAIC
Status: Not yet recruiting | Type: Observational
Sponsor: Brno University Hospital (Other)
Collaborators: Masaryk University (Other)
Responsible Party: Principal Investigator, Tereza Prokopova, MD, MD, PhD., Brno University Hospital
Other Study IDs: STRAIC
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Simulation Training; Education; Critical Care, Intensive Care; Anaesthesia
Keywords: simulation training; intensive care; European survey; education; physicians; Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study aims to describe the situation in Europe regarding simulation training during residency in Anaesthesia and Intensive Care. The main questions it aims to answer are:

How many countries in Europe have obligatory simulation training during residency? How frequent is this training? What and how is trained during simulations? How is the situation regarding funding and participation in working hours in simulation training? What are the obstacles for the countries that do not have obligatory training? Participants will fill out an electronic survey.

DETAILED DESCRIPTION:
Postgraduate education is frequently discussed in various aspects. Simulations are modern and effective tools for medical education and training during residency in Anaesthesia and Intensive Care, and are no exception. Three years ago, the survey mapped the situation of simulation-based training as an obligatory part of the residency curriculum. Now, we would like to describe the progress and identify possible factors that are preventing the further spread of simulations into postgraduate education.

ELIGIBILITY:
Inclusion Criteria:

* ESAIC NASC representatives.

Exclusion Criteria:

* not ESAIC NASC representatives.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ESAIC NASC representatives. These are clinicians representing their countries in European National Societies of Anaesthesiologists of the European Society of Anaesthesiology and Intensive Care.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
How many European countries have some type of simulation training included in the postgraduate curriculum? | 3 monts.
  This study aims to explore how many European countries have some sort of simulation included in postgraduate training. The optional or obligatory training both included.
How many European countries have obligatory simulation training in Anaesthesia and Intensive Care? | 3 months
  This study aims to explore the prevalence of obligatory simulation training in postgraduate training in Anaesthesia and Intensive Care.

SECONDARY OUTCOMES:
How extensive is the simulation training in Anaesthesiology and Intensive Care in European countries? | 3 monts
  The study aims to explore how many days of simulation training are obligatory or advised to undergo during the postgraduate training in Anaesthesia and Intensive Care.
What role does AI play in simulation training? | 3 months.
  The study aims to explore the role of AI in simulation training in Anaesthesia and Intensive Care in Europe.
Specification of simulation training | 3 months
  This study aims to describe what simulation modalities (low fidelity simulation, high fidelity simulation, etc.) are used in different European countries. Also, the themes covered by simulation training are explored.

IPD SHARING:
Plan to Share IPD: No